CLINICAL TRIAL: NCT00243802
Title: Comparison of Markers of Oxidative Stress Present in Left Atrial Appendage Tissue From Subjects With and Without Atrial Fibrillation
Brief Title: Markers of Oxidative Stress Present in Left Atrial Appendage Tissue in Patients With Atrial Fibrillation
Status: Terminated | Type: Observational
Why Stopped: Terminated.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., Principal Investigator, Emory University
Other Study IDs: 310-2005
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Inflammation
Keywords: Atrial Fibrillation; Oxidative Stress; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to look at the differences between people who have irregular heart beats coming from the upper chamber of the heart (atrial fibrillation) compared to those who do not have these irregular beats.

DETAILED DESCRIPTION:
Atrial fibrillation is an abnormal heart beat that starts in the upper parts of the heart and can cause stroke or death, if untreated. In general, treatments are not very effective with frequent relapses of the abnormal heart beats. One explanation for the high relapse rate is that the treatments might not address the underlying cause of atrial fibrillation.

Recently, we have found that atrial fibrillation is associated with increased oxidative stress in a particular part of the top parts of the heart, the left atrial appendage (LAA). Oxidative stress is a condition where abnormal oxygen forms are produced. These forms harm the cells of the heart, causing them to beat abnormally. Also, the inside of the heart becomes sticky and more likely to form blood clots. These clots, when they travel to the head, are thought to be the main cause of strokes in this condition. We have found increased oxidative stress and increased evidence of blood clotting in pig and mouse models of atrial fibrillation. We would like to see if these same findings are present in the human LAA.

In this study, we will compare blood and tissue markers of oxidative stress between patients with and without atrial fibrillation who are scheduled to undergo cardiac surgery. It is the expectation that participants with atrial fibrillation will have more abnormal markers of atrial fibrillation. This study requires participants to be seen during their routine preoperative visit, undergo a history and physical examination, give blood only once, and allow use of their discarded LAA. This tissue is routinely removed at surgery because its removal is thought to reduce the risk of strokes in patients who develop atrial fibrillation after the surgery. This happens in up to 50% of patients, thus providing the desire to remove the LAA.

ELIGIBILITY:
Inclusion Criteria:

* Cases must have atrial fibrillation documented on electrocardiographic recordings at the time of enrollment

Exclusion Criteria:

* Younger than 18 and older than 65 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and females between 18 and 65 years of age who have irregular heart beats coming from the upper chamber of the heart (atrial fibrillation).
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2005-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | 1 year
  Increased oxidative stress and increased evidence of blood clotting.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C. Dudley, Jr., M.D., Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States